CLINICAL TRIAL: NCT04874493
Title: A Pilot Study to Define PROs for Establishing a Pathway for Post Radiation or Concurrent Chemo Radiation (RT/CRT) Patient Care for Oropharyngeal Cancer
Brief Title: Patient Reported Outcome Post Radiation Therapy or Chemoradiotherapy Patient Care in Patients With Oropharyngeal Cancer
Status: Active, not recruiting | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-0015; NCI-2021-03245 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2021-0015 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2021-05-02; First posted 2021-05-05 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Oropharyngeal Carcinoma
MeSH Terms: conditions — Oropharyngeal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Observational (questionnaire): Patients complete questionnaire over 10-20 minutes at baseline, 2 times every week during weeks 1-8 of radiation therapy, and at the end of the study.
  Interventions: Other: Electronic Health Record Review; Other: Questionnaire Administration

INTERVENTIONS:
Other: Electronic Health Record Review — Review of medical records
Other: Questionnaire Administration — Complete questionnaire

SUMMARY:
This study examines patient reported outcomes post radiation therapy or chemoradiotherapy patient care in patients with oropharyngeal cancer. This study may help researchers learn about the symptoms that patients with oropharyngeal cancer have after completing radiation therapy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To provide evidence of clinically relevant symptoms for integrating into a user-friendly, automated pathway for real-time tracking and management of symptoms during post radiation therapy (RT)/chemoradiation (CRT) for oropharyngeal cancer (OPC).

OUTLINE:

Patients complete questionnaire over 10-20 minutes at baseline, 2 times every week during weeks 1-8 of radiation therapy, and at the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients who were seen for new patient evaluation at clinics and HNC centers at MD Anderson Cancer Center
* Adult patients with OPC (> 18 years old) who have been enrolled under PA14-0947

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with OPC who were seen for new patient evaluation at clinics and head and neck cancer (HNC) centers at MD Anderson Cancer Center
Sampling Method: Non-Probability Sample
Enrollment: 77 (Actual)
Dates: Start 2021-03-10 (Actual); Primary Completion 2027-02-02 (Estimated); Study Completion 2027-02-02 (Estimated)

PRIMARY OUTCOMES:
Scores of symptoms on the MD Anderson Symptom Inventory - Head and Neck (MDASI-HN) relevant to toxicities | From the end of radiation therapy (RT)/chemoradiotherapy (CRT) treatment to 2 months post-treatment
  All symptom PRO items on MDASI-HN (MD Anderson Symptom Inventory - Head and Neck (MDASI) would be rated by patients on 0 -10 of severity scale, with 0 being no symptom, and 10 being symptom as bas as imagine.

CONTACTS AND LOCATIONS:
Overall Officials: Xin S Wang, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org